CLINICAL TRIAL: NCT00319631
Title: Role of Vascular Endothelial Growth Factor (VEGF) in Acute Lung Injury/Adult Respiratory Distress Syndrome (ARDS)
Status: Withdrawn | Type: Observational
Why Stopped: Under the discretion of the PI the study has been withdrawn.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: VEGF in ARDS
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Understanding the role VEGF plays in ARDS consequently provides an ideal opportunity to discover new therapies for ARDS.

DETAILED DESCRIPTION:
In previous lab experiments, we observed evidence of pulmonary edema following alveolar epithelial overexpression of VEGF, suggesting a potential role for VEGF in ARDS. In addition, we found that preventing VEGF from reaching its target receptor(s) by overexpressing a soluble form of a VEGF receptor protein prevents edema formation.

These observations heighten the plausibility of VEGF playing an important role in the development of increased pulmonary capillary permeability during acute lung injury. Understanding this role VEGF plays in ARDS consequently provides an ideal opportunity to discover new therapies for ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that meet the American-European Consensus Conference criteria for ARDS [(1) Widespread pulmonary infiltrates; (2) Pulmonary capillary wedge pressure 18 mmHg; (3) PaOz/FiO; ratio 200; (4) compatible history], or acute lung injury [same as ARDS, but PaOz/FiOz ratio 300], or are at increased risk for developing acute lung injury because of sepsis, pancreatitis, trauma, acid aspiration, radiation or chemotherapy-induced lung toxicity, and near drowning. Pulmonary edema is divided into two broad categories: hydrostatic or cardiogenic and increased-permeability or noncardiogenic edema12. Since ARDS is noncardiogenic in origin, patients with pulmonary edema due to congestive heart failure will serve as a control group.
2. Inpatients that are endotracheally intubated.
3. Patients that are able to provide informed consent or informed consent is granted by a family member or legal health care proxy.
4. Males or females that are 18 years or older.

Exclusion Criteria:

- Individuals who are too hypoxemic for bronchoscopy to be performed safely. Patients requiring V\0z > 0.7 and/or PEEP 15 will be excluded.

2. If the patient will be unable to tolerate bronchoscopy because of severe

acidosis, tension pneumothorax, active bronchospasm, hemodynamically significant cardiac arrhythmia, or intractable shock as defined as the inability to maintain a mean arterial pressure 60 mmHg or severe uncorrectable bleeding diathesis (tendency) or as otherwise determined by the pulmonary physician.

3. Females who are pregnant will not be accepted into the study. 4. Patients with recent (48 hours) acute myocardial infraction will not be accepted into the study.

5. Patients with a history of adverse reactions to lidocaine will be not be accepted into the study. 6. Patients who lack capacity to give informed consent due to acute panic attack, "intensive care unit" psychosis or other psychologic dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects for the study will be drawn from endotracheally intubated inpatients of The New York Presbyterian Hospital-Weill Cornell Medical Center diagnosed with ALI or ARDS or who are at risk for developing ARDS.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Kaner, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided